CLINICAL TRIAL: NCT05207475
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Cerebral Amyloid Angiopathy: A Prospective, Randomized, Controlled Study
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning on Cerebral Amyloid Angiopathy. (RIC-CAA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC-CAA
Record Dates: First submitted 2021-07-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC treatment and regular treatment.
  Interventions: Device: Remote ischemic conditioning
- Regular treatment (No Intervention): Regular treatment alone.

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric auto-control device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm. The procedure will be performed twice daily for consecutive 1 years after enrollment.
  Arms: RIC group

SUMMARY:
Cerebral amyloid angiopathy (CAA) is a common form of cerebral small vessel disease, characterized by symptomatic intracerebral hemorrhage and cognitive impairment. However, no effective prevention and treatment strategies have been established. This study aims to evaluate the safety and efficacy of remote ischemic conditioning on patients with CAA.

DETAILED DESCRIPTION:
CAA is a cerebrovascular disease caused by the deposition of β-amyloid in the walls of arteries, arterioles, and capillaries in the cerebral cortex and overlying leptomeninges. It is often associated with repeated lobar intracerebral hemorrhages, progressive cognitive decline, transient neurological symptoms and gait disturbances. No treatment is specific for symptomatic management of CAA up to date. Remote ischemic conditioning is a non-invasive strategy to protect the brain. The clinical trials have demonstrated that daily limb RIC seems to be potentially effective in patients with cerebral small-vessel disease in slowing cognition decline and reducing white matter hyperintensities. Thereby, investigators design this study to assess whether RIC has a beneficial effect on CAA.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥55 and ≤85.
2. The diagnosis of probable CAA and probable CAA with supporting pathology by the Boston criteria.
3. Signed and dated informed consented is obtained.

Exclusion Criteria:

1. Familial hereditary CAA or other hereditary small-vessel disorders.
2. Previous intracranial hemorrhage caused by other reasons, such as tumor, cerebral cavernous angioma, ruptured aneurysm, arteriovenous malformation, venous sinus thrombosis and so on.
3. A history of stroke within 3 months.
4. The degree of intracranial or extracranial large artery stenosis >50%.
5. Clinical diagnosis of probable AD by National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
6. Significant cognitive impairment (defined as Mini-mental State Examination (MMSE) score of ≥20 (primary school) or ≥24 (junior school or above) or other diseases resulting from severe cognitive impairment.
7. Inability to walk 6m unaided or other conditions that affected gait performance, such as Parkinson.
8. Illiteracy and patients with severe visual or hearing impairment.
9. Contraindication to MRI scan, such as intracranial metal implants, cardiac pacemaker, severe claustrophobia, history of seizures and so on.
10. Patients with missing or poor-quality MRI sequences at baseline and follow-up.
11. Patients with a pre-existing neurological deficits (modified Ranks scale score >2) or psychiatric disease that would confound the neurological or functional evaluations.
12. Alcohol dependence and other psychoactive substance abuse
13. Contraindication for remote ischemic conditioning: severe soft tissue injury, limb deformities, fracture, atrial fibrillation or peripheral vascular disease in the upper limbs.
14. Life expectancy of less than 1 year due to co-morbid conditions.
15. Severe, sustained hypertension (SBP > 180 mmHg or DBP > 110 mmHg).
16. Severe renal or hepatic disease.
17. Known pregnancy (or positive pregnancy test), or breast-feeding.
18. Concurrent participation in another research protocol for investigation of another experimental therapy.
19. Any condition which, in the judgment of the investigator, might increase the risk to the patient.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Changes of volume of WMHs. | From baseline to 6 months and 1 year treatment.
  The volume of WMHs was measured on Flairs at 6months and 12months.

SECONDARY OUTCOMES:
Adverse events related to RIC treatment. | From baseline to 6 months and 1 year treatment.
  Adverse events related to RIC treatment, such as mucocutaneous hemorrhage, changes in coagulation function and so on.
Incidence of cardio-cerebral vascular events. | From baseline to 6 months and 1 year treatment.
  Incidence of cardiovascular and cerebrovascular events,such as Intracranial hemorrhage, subarachnoid hemorrhage, CAA-related transient focal neurological episodes（CAA-TFNEs）, CAA-related Inflammation（CAA-ri），ischemic stroke during follow-up.
Changes of the cerebral blood flow in MRI ASL. | From baseline to 6 months and 1 year treatment.
  Changes of the CBF are assessed by Arterial Spin Labeling (ASL) MRI techniques at 6months and 12months.
Changes of cognition evaluation on MoCA. | From baseline to 6 months and 1 year treatment.
  We used MoCA to evaluate the cognitive functions,of subjects at 6months and 12months, such as memory, execution, visuospatial function and so on.
Changes of cognition evaluation on TMT tests. | From baseline to 6 months and 1 year treatment.
  We used TMT tests to evaluate execution and and so on at 6months and 12months.
Changes of cognition evaluation on stroop tests. | From baseline to 6 months and 1 year treatment.
  We used stroop tests to evaluate execution and and so on at 6months and 12months.
Changes in evaluation of Timed-Up-and-Go tests. | From baseline to 6 months and 1 year treatment.
  We used Timed-Up-and-Go tests to evaluate the gait function of subjects at 6months and 12months.
Changes of the whole volume of microbleeds. | From baseline to 6 months and 1 year treatment.
  The volume of microbleeds was measured on QSM at 6months and 12months.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490
- [Background] Chen SJ, Tsai HH, Tsai LK, Tang SC, Lee BC, Liu HM, Yen RF, Jeng JS. Advances in cerebral amyloid angiopathy imaging. Ther Adv Neurol Disord. 2019 May 3;12:1756286419844113. doi: 10.1177/1756286419844113. eCollection 2019. PMID 31105769